CLINICAL TRIAL: NCT02331082
Title: Integrating Pediatric Care Delivery in Rural Healthcare Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Possible (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: hssnyaya
Record Dates: First submitted 2013-08-08; First posted 2015-01-06 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Infant Mortality; Under-two Mortality
Keywords: Infant Mortality; Under-two mortality; Maternal Mortality; Implementation Research; Health Systems Strengthening; Chronic Disease Management; Commuity Health Workers
MeSH Terms: conditions — Infant Death; Maternal Death | interventions — Chronic Care Model; Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Existing healthcare system
  Interventions: Other: Existing healthcare system
- Health System Improvement (Experimental): Structured Quality Improvement Chronic Care Model Integrated Electronic Medical Record Solar-powered electrical supply Performance-based financing
  Interventions: Other: Structured Quality Improvement; Other: Chronic Care Model; Device: Integrated Electronic Medical Record; Device: Solar-powered electrical supply; Behavioral: Performance-based financing

INTERVENTIONS:
Other: Structured Quality Improvement — For structured quality improvement, trained healthcare providers (primarily doctors from referral hospital) will serve as mentors to mid-level providers. The mentors will facilitate on-site trainings of primary care with mid-level providers at the district hospital. Mentors will also travel monthly to the healthcare facilities themselves to provide training both in the direct context of clinical care and to provide feedback based upon surveillance and monitoring data. The focus will be on the techniques from the Institute for Healthcare Improvement's Model for Improvement, including Plan-Do-Study-Act cycles, run charts, and root cause analyses. Finally, they will work with the clinical healthcare staff to identify resource needs from the local government for maintenance, water, electricity, and supplies. These resource needs will be addressed through an integrated supply chain management system across the tiers of the healthcare system.
  Other Names: Clincal Mentorship; Supply Chain Management
  Arms: Health System Improvement
Other: Chronic Care Model — Senior physicians trained in mentorship of non-physician mid-level providers will provide decision support for mid-level providers in the current district healthcare system with specific protocols for target conditions. We will add the following elements: focus on mid-level, non-physician providers as the primary clinicians within the intervention; intensive Community Health Worker (CHW) outreach for detection, screening, follow-up of patients, and encouragement of patient self-care and behavior change; and focused effort on the seamless care coordination of patients across the tiers of the system. Through trainings of CHWs, much of patient self-management comes in the form of home visits that reinforce clinic and hospital counseling, including risk management and prevention. CHWs will be trained in the counseling of each target condition, with counseling largely occurring in the patients' homes, where much of the challenges of chronic disease management and behavior change lie.
  Other Names: Task-Shifting; Healthcare Systems Strengthening
  Arms: Health System Improvement
Device: Integrated Electronic Medical Record — Clinical information systems. We are developing a system for tracking patients that integrates across each of the tiers using an electronic medical record. This is a key technology in supporting each of the above delivery system design elements.
  Other Names: Electronic Medical Record
  Arms: Health System Improvement
Device: Solar-powered electrical supply — As a component of our comprehensive healthcare systems strengthening intervention, we are installing solar panels at community-level clinics to ensure continuous electrical supply for medical devices and technology.
  Other Names: Solar Panel
  Arms: Health System Improvement
Behavioral: Performance-based financing — As part of our healthcare systems strengthening intervention, we have established a performance-based financing agreement with the Government of Nepal that conditionally funds healthcare delivery based on population-level health outcomes and quality healthcare service delivery. In this arrangement, the Government serves as a regulator of healthcare delivery rather than a primary provider of healthcare services.
  Arms: Health System Improvement
Other: Existing healthcare system — This is the current rural, district-level public sector healthcare infrastructure of rural Nepal that is not strengthened during the study.
  Other Names: Control
  Arms: Control

SUMMARY:
Globally, over seven million children under the age of five die each year, although a suite of interventions-safe delivery care, neonatal care and resuscitation, and management of childhood diarrhea, malnutrition, and pneumonia-can prevent many of these deaths when implemented within functioning health systems. This study will include a quasi experimental, stepped wedge, cluster-controlled trial of a mobile health care coordination and quality improvement intervention designed to facilitate comprehensive health systems strengthening. It will do this through training and equipping community-level health care clinics to manage chronic diseases through use of the Chronic Care Model, structured quality improvement sessions to promote clinical mentorship, and use of an integrated electronic medical record to provide real-time data for disease surveillance. The investigators hypothesize that improving upon the health system in these ways will lead to a 25% reduction in under-two mortality through improved services for the citizens of Achham, Nepal.

DETAILED DESCRIPTION:
Introduction: A central challenge in the delivery of evidence-based interventions to promote under-five child survival is the coordination of care across the multiple tiers of the health system, from frontline health workers, to primary care clinics, to district hospitals, to specialty providers. Additionally, children who survive or avoid once-fatal diseases such as congenital and rheumatic heart diseases, prematurity, neurodevelopmental conditions, and disabilities sustained from traumatic injuries, are increasingly living well into adolescence, young adulthood, and beyond. Healthcare delivery systems in resource-limited settings, however, are ill-equipped to manage such patients' care. Mobile technologies, coupled with effective management strategies, may enhance implementation and coordination of evidence-based interventions, but few controlled trials exist to validate this. Particularly lacking are strategies that incorporate mobile technologies in an integrated manner across the health system.

Intervention: We have developed a mobile health care coordination and quality improvement intervention within two rural district healthcare systems in Nepal, where the child mortality rate is an estimated 82 per 1,000, and coordination of child health care is poor. Firstly, the intervention aims to increase the timely engagement in acute care for children under the age of five to receive evidence-based World Health Organization protocols aimed at reducing child mortality-Integrated Management of Pregnancy and Childbirth, Integrated Management of Childhood Illness, Integrated Management of Emergency and Essential Surgical Care, and Community-based Management of Severe Acute Malnutrition. Secondly, the intervention aims to implement a Chronic Care Model for pediatric patients under the age of twenty suffering from a chronic disease (congenital and rheumatic heart disease, diabetes, depression, epilepsy, asthma, musculoskeletal and neurodevelopmental disabilities, and pre- and post-surgical conditions).

Analysis: We will conduct a quasi-experimental, stepped-wedge, cluster-controlled trial. The primary outcome of this trial will be under-two mortality. We hypothesize a 25% reduction in under-two mortality rate during the intervention periods, relative to the control period. We hypothesize a 50% improvement in follow-up rates, a 30% improvement in global symptoms score, a 20% reduction in disability score, and a 20% reduction in inpatient days in hospital. We will use both quantitative and qualitative methods to assess the scalability of the intervention in terms of logistics, human resources, costs, and utilization.

Impact: Rigorous evaluations of systems-level child healthcare interventions are needed to drive global healthcare policies and their implementation. The trial proposed here will inform the potential impact and scalability of health systems strengthening interventions.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Reproductive age, 15-49 years
* Resides within 14 village clusters that comprise experimental/control arms

Exclusion Criteria:

* n/a

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7000 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Under-two mortality rate | Five years
  We expect the intervention will lead to a 25% decrease in under-two mortality in the experimental arm.
Infant mortality rate | Five years
  We expect the intervention will lead to a 25% decrease in the infant mortality rate in the experimental arm.
Neonatal mortality rate | Five years
  We expect the intervention will lead to a 25% decrease in the neonatal mortality rate in the experimental arm.

SECONDARY OUTCOMES:
Institutional Birth Rate | Five years
  We expect the intervention will lead to a 25% increase in Institutional Birth Rate among reproductive-age women in the experimental arm.
Antenatal Care Completion Percentage | Five years
  We expect the intervention will lead to a 25% increase in number of pregnant women completing all 4 antenatal care visits in the experimental arm.
Postpartum contraceptive prevalence rate | Five years
  We expect the intervention will lead to a 20% increase in postpartum contraceptive prevalence rate among reproductive age women who have delivered in the past 2 years in the experimental arm.
Preterm delivery rate | Five years
  We expect the intervention will lead to 25% fewer preterm births in the experimental arm.
Low birthweight delivery rates | Five years
  We expect the intervention will lead to a 25% reduction in babies born with low birthweights in the experimental arm
Percentage of stillbirths | Five years
  We expect the intervention will lead to 25% fewer stillbirths in the experimental arm.

CONTACTS AND LOCATIONS:
Overall Officials: David Citrin, PhD, MPH, Study Director — Possible; Biraj Karmacharya, MBBS, MSc, Study Chair — University of Washington
Locations (2):
- Nepal (2):
  - Bayalpata Hospital, Sanfebagar, Achham
  - Charikot Primary Health Center, Bhimeshwor, Dolakha

REFERENCES:
- See also: Possible — http://possiblehealth.org/
- See also: Healthcare Systems Design Group — http://hsdg.partners.org/